CLINICAL TRIAL: NCT05362799
Title: Different Induction Protocols in PCOS After Clomiphene Citrate Failed Pregnancy in Non-IVF Cycles
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Mohamed Maher, Professor, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3/2022/OBG
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Letrozole; lactitol; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- GROUP 1 (Active Comparator): GROUP 1: Participants of this group will receive Letrozol (Femara, Novartis) at a dose of 2.5mg twice daily starting from day 3 of the cycle for 5 days.
  Interventions: Drug: Letrozol (Femara, Novartis)
- GROUP 2 (Active Comparator): GROUP 2: Participants of this group will receive Letrozol (Femara, Novartis) at a dose of 2.5mg twice daily starting from day 3 of the cycle for 5 days. Metformin (Cidophage 500 mg, Cid Pharmaceuticals, Egypt) 500 mg twice daily will also started from day 3 till the date of doing pregnancy test
  Interventions: Drug: Letrozol (Femara, Novartis) combined with Metformin (Cidophage 500 mg, Cid Pharmaceuticals, Egypt)
- GROUP 3 (Active Comparator): Participants of this group will receive highly purified lyophilized Uroffollitropin (Fostimon, IBSA Institut Biochimique SA, Lugano, Switzerland.) at a dose of 75IU S.C or IM starting from day 3 of the cycle for 5 days. Readjustment of the dose will occur upon the results of day 8 folliculometry.
  Interventions: Drug: highly purified lyophilized Uroffollitropin (Fostimon, IBSA Institut Biochimique SA, Lugano, Switzerland)
- GROUP 4 (Active Comparator): Participants of this group will receive highly purified lyophilized Uroffollitropin (Fostimon, IBSA Institut Biochimique SA, Lugano, Switzerland.) at a dose of 75IU S.C or IM starting from day 3 of the cycle for 5 days. Readjustment of the dose will occur upon the results of day 8 folliculometry. Metformin (Cidophage 500 mg, Cid Pharmaceuticals, Egypt) 500 mg twice daily will also started from day 3 till the date of doing pregnancy test
  Interventions: Drug: highly purified lyophilized Uroffollitropin (Fostimon, IBSA Institut Biochimique SA, Lugano, Switzerland) combined with metformin

INTERVENTIONS:
Drug: Letrozol (Femara, Novartis) — Letrozol (Femara, Novartis) at a dose of 2.5mg twice daily starting from day 3 of the cycle for 5 days.
  Arms: GROUP 1
Drug: Letrozol (Femara, Novartis) combined with Metformin (Cidophage 500 mg, Cid Pharmaceuticals, Egypt) — Participants of this group will receive Letrozol (Femara, Novartis) at a dose of 2.5mg twice daily starting from day 3 of the cycle for 5 days. Metformin (Cidophage 500 mg, Cid Pharmaceuticals, Egypt) 500 mg twice daily will also started from day 3 till the date of doing pregnancy test
  Arms: GROUP 2
Drug: highly purified lyophilized Uroffollitropin (Fostimon, IBSA Institut Biochimique SA, Lugano, Switzerland) — Participants of this group will receive highly purified lyophilized Uroffollitropin (Fostimon, IBSA Institut Biochimique SA, Lugano, Switzerland) at a dose of 75IU S.C or IM starting from day 3 of the cycle for 5 days. Readjustment of the dose will occur upon the results of day 8 folliculometry.
  Arms: GROUP 3
Drug: highly purified lyophilized Uroffollitropin (Fostimon, IBSA Institut Biochimique SA, Lugano, Switzerland) combined with metformin — Participants of this group will receive highly purified lyophilized Uroffollitropin (Fostimon, IBSA Institut Biochimique SA, Lugano, Switzerland.) at a dose of 75IU S.C or IM starting from day 3 of the cycle for 5 days. Readjustment of the dose will occur upon the results of day 8 folliculometry. Metformin (Cidophage 500 mg, Cid Pharmaceuticals, Egypt) 500 mg twice daily will also started from day 3 till the date of doing pregnancy test
  Arms: GROUP 4

SUMMARY:
The aim of this study will be to compare between 4 different induction protocols in women who:

1. Failed to achieve ovulation after clomiphene citrate treatment at a dose of 150mg daily (if the patient can tolerate this dose) for 5 days for 3 cycles or only 100 mg daily for the same duration (if she can't tolerate higher dose)
2. Failed to achieve pregnancy after 3 cycles of ultrasound indicated ovulation with clomiphene citrate treatment at a dose of 100mg or 150mg daily.

All induction protocols will be carried out in non-IVF cycles, and continued for 3 cycles or until pregnancy whichever will be earlier.

DETAILED DESCRIPTION:
The study will include 4 treatment groups:

GROUP 1: Participants of this group will receive Letrozol (Femara, Novartis) at a dose of 2.5mg twice daily starting from day 3 of the cycle for 5 days.

GROUP 2: Participants of this group will receive Letrozol (Femara, Novartis) at a dose of 2.5mg twice daily starting from day 3 of the cycle for 5 days. Metformin (Cidophage 500 mg, Cid Pharmaceuticals, Egypt) 500 mg twice daily will also started from day 3 till the date of doing pregnancy test GROUP 3: Participants of this group will receive highly purified lyophilized Uroffollitropin (Fostimon, IBSA Institut Biochimique SA, Lugano, Switzerland.) at a dose of 75IU S.C or IM starting from day 3 of the cycle for 5 days. Readjustment of the dose will occur upon the results of day 8 folliculometry.

GROUP 4: Participants of this group will receive highly purified lyophilized Uroffollitropin (Fostimon, IBSA Institut Biochimique SA, Lugano, Switzerland.) at a dose of 75IU S.C or IM starting from day 3 of the cycle for 5 days. Readjustment of the dose will occur upon the results of day 8 folliculometry. Metformin (Cidophage 500 mg, Cid Pharmaceuticals, Egypt) 500 mg twice daily will also started from day 3 till the date of doing pregnancy test For follow up:US folliculometry will be done on Day 8 in all groups. Further appointments for folliculometry will be given upon the response. Dominant follicle will be diagnosed on Day 8 if the average follicular diameter is 12mm or more (taken in 2 perpendicular diameters) then follow up will be continued till the diameter reaching 18-22mm so that triggering ovulation will be carried out by administration of human chorionic gonadotrophins (Epifasi 5000 IU, ampoule, EIPICO pharmaceuticals, Egypt). All women will be advised to receive the injection within 12 hours of the last follicular measurement. Women will be advised to have unprotected intercourse 24-36h following hCG injection. Serum β-hCG will be measured after 2 weeks to check for pregnancy and US will be performed after 2-4 weeks from B-hCG results to confirm the presence of pregnancy.

Each couple will be involved in the study for 3 treatment cycles if pregnancy will not occur but still having the option not to continue in our study where we will manage them outside the study protocol.

Women who will get pregnant will be followed for 12w gestational age for possible detection of 1st trimester abortion.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged between 20-35 years
2. Body mass index ≤ 30
3. Primary or secondary infertility for ≥1 year due to PCOS (diagnosed based on Rotterdam criteria which require the presence of two of the following: Oligo\an ovulation , hyperandrogenism, polycystic ovaries on ultrasound)
4. Failure to achieve ovulation after clomiphene citrate treatment at a dose of 150mg daily (if the patient can tolerate this dose) for 5 days for 3 cycles or only 100 mg daily for the same duration (if she can't tolerate higher dose)
5. Failure to achieve pregnancy after 3 cycles of ultrasound indicated ovulation with clomiphene citrate treatment at a dose of 100mg or 150mg daily.
6. Day-2 follicle-stimulating hormone less than 12 IU/ml
7. Normal serum prolactin and thyroid function
8. Normal uterine cavity
9. At least one patent tube
10. Male partner with normal semen count and motility according to WHO criteria

Exclusion Criteria:

1. Male factor infertility
2. Bilateral tubal block
3. Uncontrolled thyroid dysfunction
4. Uterine factor of infertility.
5. Known cases with endometriosis.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of ovulation | 18 month
  US detection of one or more follicles of 18mm or more
Number of dominant follicles | 18 month
  US detection of follicles >18mm
Endometrial thickness | 18 months
  US assessment of endometrial thickness

SECONDARY OUTCOMES:
Occurrence of pregnancy which will be subdivided into: chemical pregnancy or clinical pregnancy | 18 months
  type of pregnancy
Total number of patients getting pregnant after each treatment cycle in each group | 18 months
  record occurrence of pregnancy
Number of cycles cancelled in each group | 18 months
  detect cycle cancellation
Number of patients developing OHSS in each group | 18 months
  detect ovarian hyperstimulation syndrom
Number of patients having multiple pregnancy in each group | 18 months
  detect multiple pregnancy
Number of patients ended by 1st trimester miscarriage in each group | 18 months
  detect miscarriage
Side effects recorded in each group | 18 months
  record side effects that patients complaint

IPD SHARING:
Plan to Share IPD: No